CLINICAL TRIAL: NCT02232490
Title: Phase III Randomized, Placebo-controlled Clinical Trial of Hepcortespenlisimut-L (Hepko-V5) Versus Placebo in Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Liver Cancer Immunotherapy: Placebo-controlled Clinical Trial of Hepcortespenlisimut-L
Acronym: Hepko-V5
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Responsible Party: Principal Investigator, Aldar Bourinbaiar, Investigator, Immunitor LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Immunitor Hepko-V5; IMM05 (Other: Immunitor)
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma; HCC; Liver Cancer
Keywords: AFP; alpha-fetoprotein; cancer vaccine; cirrhosis; hepatitis; HCC; hepatocellular carcinoma; immunotherapy; liver tumor; Cholangiocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Fibrosis; Hepatitis; Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hepcortespenlisimut-L (Experimental): Experimental placebo-controlled clinical of hepcortespenlisimut-L (V5) therapeutic vaccine against HCC
  Interventions: Biological: hepcortespenlisimut-L
- placebo (Placebo Comparator): placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: hepcortespenlisimut-L — hepcortespenlisimut-L (V5) is given in experimental arm
  Other Names: V5
  Arms: hepcortespenlisimut-L
Biological: Placebo
  Arms: placebo

SUMMARY:
Phase III, randomized, placebo-controlled, double-blinded trial aimed to seek the therapeutic benefit of hepcortespenlisimut-L (Hepko-V5) in subjects with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Phase III, randomized, placebo-controlled, double-blinded trial aimed to seek the therapeutic benefit of hepcortespenlisimut-L (Hepko-V5) in subjects with advanced hepatocellular carcinoma. The results will be compared to placebo. The trial duration is 3 months and will consist of one stage with baseline laboratory evaluation including AFP levels with follow-up at monthly intervals. In addition pre-entry abdominal CT scan and end-study CT scan will be preformed. The clinical evaluation will be quantified according to special performance questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Subjects who are at least 18 years old and are willing and capable of providing informed consent. Both men and non-pregnant women will be included.

HCC diagnosis documented prior to Study Entry by either cytology/histology, CT scan, and AFP serum test higher or equal to 30 IU/ml.

All subjects with reproductive potential are advised to utilize effective contraception throughout the course of this study.

Health score status at baseline. Agreement to participate in the study and to give at least 3 samples of blood for lab tests.

Readily available home or o other address where patient can be found. -

Exclusion Criteria:

Subjects who might have already taken V5 in prior trials and have no baseline data. Those who met inclusion criteria can be retrospectively enrolled. Pregnant or breast-feeding women are excluded.

Subjects who have taken other immunomodulatory therapies within 2 months prior to Entry: systemic corticosteroids, immune globulin (IV gamma globulin, IVIG), interferons, interleukins, pentoxifylline (Trental), thalidomide, filgrastim (G-CSF), sargramostim (GM-CSF); dinitrochlorobenzene (DNCB), thymosin alpha 1 (thymosin alpha), thymopentin, inosiplex (Isoprinosine), polyribonucleoside (Ampligen), ditiocarb sodium (Imuthiol), any locally available immune modulators, and any other therapeutic or preventive HCC vaccine. Subjects requiring concurrent participation in another experimental research treatment study, or who received an experimental agent within four weeks prior to Study Entry.

Evidence of active or acute cardiac disease, epilepsy, or life-threatening diseases unrelated to HCC.

Medical conditions such as active alcohol or substance abuse, or psychological issues that in the opinion of the local investigator would interfere with adherence to the requirements of this study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
changes in plasma AFP | 3 months
  Changes in plasma AFP levels at monthly intervals

SECONDARY OUTCOMES:
CT scan | 3 months
  changes in tumor size/mumber at 3 months compared to baseline

OTHER OUTCOMES:
adverse effects | 3 months
  evaluation of adverse effects if any

CONTACTS AND LOCATIONS:
Overall Officials: aldar bourinbaiar, Study Director — Immunitor LLC
Locations (1):
- Immunitor LLC, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: Yes
DATA TO BE SHARED WITH COLLABORATORS

REFERENCES:
- See also: Interim Phase II trial outcome — http://www.prweb.com/releases/2014/06/prweb11965485.htm
- See also: Phase II results abstract — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4649454/